CLINICAL TRIAL: NCT00792441
Title: Effect of Specific Inspiratory Inspiratory Training(SIMT)in the Patients With Ventilatory Dependence on Lung Function and Weaning Outcomes
Brief Title: Specific Inspiratory Muscle Training (SIMT)in the Patients With Ventilatory Dependence
Acronym: SIMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saikaew Chuachan (Other)
Collaborators: Khon Kaen University (Other)
Responsible Party: Sponsor-Investigator, Saikaew Chuachan, Associated Medical Science, Khon Kaen University
Organization: Khon Kaen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KKU4950900071; HE501034 (Other: KKU)
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Ventilatory Defect
Keywords: Specific inspiratory muscle training(SIMT); Loaded deep breathing; Weaning; Mechanical ventilation; Respiratory muscle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention group (No Intervention): Patients with mechanical ventilated who met the criteria for weaning from medical doctor in Srinagarind hospital, Khon Kaen University
  Interventions: Device: intervention group

INTERVENTIONS:
Device: intervention group — inspiratory muscle training at 50% of peak negative inspiratory muscle training (PNIP)will be performed with 6 breathe/set, 10 set/day, once a day for 28 days.
  Other Names: BreatheMax v.1; water pressure threshold breathing (WPTB)

SUMMARY:
Prolong mechanical ventilation cause to respiratory muscle weakness and high risk to weaning failure,the investigators hypothesize that

1. Specific inspiratory muscle training (SIMT) using threshold loaded breathing device (BreatheMAX V.1)in patients with ventilator dependence will improve inspiratory muscle strength
2. SIMT will improve lung function in patients with ventilatory dependence.
3. SIMT will improve weaning success in patients with ventilatory dependence.

DETAILED DESCRIPTION:
Prolonged mechanical ventilation cause detrimental effects on lung function and high risk of lung complications and standard weaning protocols are not successful in a number of patients. The strength of the inspiratory muscles is important factors in the success of weaning. Although, the inspiratory muscles are trained by manipulating the ventilator sensitivity and made of ventilation in the traditional protocol, the muscle function might not improved sufficiently to sustain independent and spontaneous breathing. Consequently, specific inspiratory muscle training is indicated and has been studied in patient with weaning failure. However, there is little evidence available and no firm conclusion can be drown. Therefore, the purpose of this study is to determine whether specific IMT training using the local made loaded threshold IMT device can improve lung function and accelerate the weaning process.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have been mechanically ventilated > 72 hours and start to weaning from medical order or ventilator dependent patients who have failed to wean prior to study.
* Normal arterial blood gas (PaCO2 < 50mmHg, PaO2 > 60 mmHg on FiO2 <0.5 or SaO2 > 90%, PH 7.35-7.45).
* Cardiovascular stability (HR ≤ 140 beats/min, systolic BP 90-140 mmHg and diastolic BP 60-90 mmHg, with no or minimal vasopressors)
* Good consciousness, cooperation and can sit in an upright position > 30 minutes

Exclusion Criteria:

* Persistent homodynamic instability.
* Severe breathlessness at rest when spontaneous breathing.
* Coronary heart disease with angina.
* Life threatening arrhythmia (VF, VT).
* Sedation Ramsay scale > 2
* Severity of disease APACHE II score > 29

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Peak Negative Inspiratory Pressure (PNIP) | every 7 day for 28 days

SECONDARY OUTCOMES:
Lung compliance | every 7 day for 28 days
Vital capacity | every 7 day for 28 days
Rate perceived breathlessness | every 7 day for 28 day
Airway resistance | every 7 day for 28 days.
Tidal volume | every 7 day for 28 days.
Minute ventilation | every 7 day for 28 days.
End tidal carbondioxide (PetCO2) | every 7 day for 28 days.
SpO2 | every 7 day for 28 days.
Heart rate | every 7 day for 28 days.
Respiratory rate | every 7 day for 28 days.
Weaning success | every 7 day for 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Reechaipichitkul Wipa, MD, Study Director — Department of medicine, Faculty of medicine, Khon Kaen university; Chulee CU Jones, Philosophy, Study Director — Physical Therapy department, Faculty of Associated Medical Sciences, Khon Kaen university; Saikaew Chuachan, Bachelor, Study Chair — Physical Therapy department, Faculty of Associated Medical Sciences, Khon Kaen university
Locations (1):
- Respiratory Intensive Care Unit (RICU),Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen, Thailand